CLINICAL TRIAL: NCT05775549
Title: FLAME - First Line olAparib Maintenance bEyond BRCA An Observational Cohort Study to Characterize the Outcomes of Olaparib Maintenance Monotherapy Beyond BRCA Mutant Status in Newly Diagnosed Advanced Ovarian Cancer
Brief Title: A Study to Characterize the Outcomes of Olaparib Maintenance Monotherapy in Newly Diagnosed BRCAwt Ovarian Cancer
Acronym: FLAME
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: D0818R00008
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Advanced Ovarian Cancer
Keywords: Real-world evidence; Homologous recombination deficiency; breast cancer gene; breast cancer gene mutated; breast cancer gene wild type
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Patients with newly diagnosed AOC BRCAwt with known HRD status who have been prescribed 1L olaparib maintenance treatment.
  Interventions: Other: None (Observational Study)

INTERVENTIONS:
Other: None (Observational Study) — Not Applicable since observational study
  Other Names: Observational Study

SUMMARY:
This study will collect the data from existing patient medical records at US cancer centers. The study will include patients with BRCAwt ovarian cancer who have been prescribed first line (1L) olaparib maintenance treatment.

DETAILED DESCRIPTION:
This is a United States (US) based multicenter, retrospective, observational cohort study with data abstracted from patient medical records.

In this observational study, it is planned to include approximately 150 US female patients with newly diagnosed advanced ovarian cancer (AOC) who were tumor biomarker tested between first diagnosis with AOC and first prescription of 1L olaparib maintenance monotherapy as tumor breast cancer gene wild type (BRCAwt) with a known homologous recombination deficiency (HRD) status.

This retrospective cohort study will include patients with first olaparib prescription between Jan 2017 and Dec 2021. All data collection will be retrospective. Data will be collected from the date of first olaparib prescription (index date) with a follow-up period of at least 18 months post index date.

ELIGIBILITY:
Inclusion Criteria:

* Female adult, age ≥ 18 years
* BRCAwt AOC diagnosed with any approved BRCA test
* Has documented HRD status based on available test results
* Received 1L olaparib maintenance monotherapy following platinum chemotherapy
* Patients must have been treated with platinum-based chemotherapy at first-line

Exclusion Criteria:

* Received another poly adenosine diphosphate ribose polymerase (PARP) inhibitor or bevacizumab before or while prescribed olaparib
* Participation in an interventional clinical study

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed AOC BRCAwt with available HRD status who have been prescribed 1L olaparib maintenance treatment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Clinical and Demographics characteristics | At Index date - first olaparib prescription (Jan 2017 to Dec 2021)
  Clinical and Demographic characteristics including disease/FIGO stage, histology and tumor grade at initial Ovarian Cancer diagnosis, cancer antigen 125 (CA-125) level, Eastern Cooperative Oncology Group (ECOG) or other performance status, number and type of chemotherapy cycles, cytoreductive/debulking surgery type and outcomes, and selected comorbidities at index date will be described.
  Summary statistics will be used to describe the Demographics and clinical characteristics.
  The outcome will be measured for HRD+ patients.

SECONDARY OUTCOMES:
Real-world time to first subsequent treatment or death (rwTFST) | Jan 2017 to Jun 2023
  rwTFST is defined as the time from the index date (date of the first olaparib prescription) to the earliest of the date of death or commencement of first subsequent anticancer treatment.
  The outcome will be measured for HRD+ patients.
Real-world time to treatment discontinuation or death (rwTTD) | Jan 2017 to Jun 2023
  rwTTD is defined as the time from the index date to the earliest of the date of death or discontinuation of olaparib.
  The outcome will be measured for HRD+ patients.
Number of patients with clinical event of interest (CEI) | Jan 2017 to Jun 2023
  To summarize the real-world safety and tolerability profile based on pre-specified CEIs of 1L olaparib maintenance monotherapy in BRCAwt newly diagnosed AOC patients regardless of HRD status.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Tampa, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0818R00008&attachmentIdentifier=e02baacb-9e72-41f9-b1aa-fe69ba20ec44&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=